CLINICAL TRIAL: NCT01661855
Title: A Pilot Study of Riluzole vs. Placebo in the Treatment of Children and Adolescents With Autism Spectrum Disorders
Brief Title: A Pilot Study of Riluzole Versus Placebo in the Treatment of Children and Adolescents With ASD
Acronym: RILISE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Holland Bloorview Kids Rehabilitation Hospital (Other)
Collaborators: McMaster University (Other); The Hospital for Sick Children (Other); The University of Western Ontario (Unknown); Unity Health Toronto (Other); University of Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RILISE-07-2013
Record Dates: First submitted 2012-07-26; First posted 2012-08-10 (Estimated); Last update posted 2025-07-16 (Actual); Status verified 2017-03

CONDITIONS: Autism Spectrum Disorders
Keywords: Autism Spectrum Disorders
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Riluzole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Riluzole (Active Comparator)
  Interventions: Drug: Riluzole
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Riluzole — 50mg once daily (QD) for 12 weeks for participants 6-11 years old; 50mg twice daily (BID) for 12 weeks for participants 12-17 years old
  Other Names: Rilutek
  Arms: Riluzole
Drug: Placebo — Placebo comparator once daily (QD) for 12 weeks for participants 6-11 years old; Placebo comparator twice daily (BID) for 12 weeks for participants 12-17 years old
  Arms: Placebo

SUMMARY:
This study will examine the potential efficacy and safety of riluzole for core and associated symptom domains of autism and will explore biological markers of safety and treatment response.

DETAILED DESCRIPTION:
There are no pharmacologic treatments available for social function deficits in individuals with Autism Spectrum Disorders (ASD). The data for pharmacologic treatment of repetitive behaviors in this disorder has also become difficult to interpret given that the last two large multisite trials of selective serotonin reuptake inhibitors (SSRIs) in autism are reported to be negative for the treatment of repetitive behaviors. Only the associated symptom of irritability has 2 drugs with FDA indications whereas no systematic data exists on the pharmacologic treatment of anxiety in ASD, and response to rates to stimulants for hyperactivity are lower than what is seen in attention deficit hyperactivity disorder (ADHD). In addition, there are no biological markers of treatment response identified in this population at this point. This study will examine the potential efficacy and safety of riluzole for core and associated symptom domains of autism and will explore biological markers of safety and treatment response.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female outpatients 6-17 years of age inclusive, with a mental age equivalent ≥ 18 months at Screening visit.
2. Meet Diagnostic and Statistical Manual (DSM-IV) criteria for an ASD.
3. Have a Clinician's Global Impression-Severity (CGI-S) score ≥ 4 (moderately ill) at Screening.
4. If already receiving stable interventions must meet the following criteria:

   1. If already receiving stable concomitant medications affecting behavior, must be on a stable dose during the preceding 1 month prior to Screening (with the exception of fluoxetine, where a period of 6 weeks is needed), and will not electively initiate new or modify ongoing medications for study duration.
   2. If already receiving stable non-pharmacological educational, behavioral, and/or dietary interventions, have continuous participation during the preceding 3 months prior to Screening, and not electively initiate new or modify ongoing interventions for the duration of the study.
5. Have normal physical examination and laboratory test results at Screening. If abnormal, the finding(s) must be deemed clinically insignificant by the Investigator.
6. Ability to complete assessments- fluency in English (parent; patient, if verbal).
7. Consent to participate in the Province of Ontario Neurodevelopmental (POND) study and commitment to completing as many stages as possible of the phenotyping measures (Stages 1, 2 and 3), genomics component, and interest in being imaged through POND.
8. Ability to obtain written informed consent from the participant, if developmentally appropriate. If a participant does not have the capacity to consent, ability to obtain assent (if developmentally appropriate), as well as written informed consent from their parent(s)/legal guardian.

Exclusion Criteria:

1. Pregnant female patients; sexually active female patients on inadequate birth control.
2. Patients with a serious medical condition that, based on Investigator judgment, might interfere with the conduct of the study, confound interpretation of the study results, or endanger their own well-being. Patients with evidence or history of malignancy or any significant hematological, endocrine, cardiovascular (including any rhythm disorder), respiratory, renal, hepatic, or gastrointestinal disease, not including mild common pediatric diseases in these areas that are stable (e.g. mild asthma, constipation, etc.).
3. Patients with unstable epilepsy (i.e. seizures occurring within the last 6 months), or patients with epilepsy who are not on stable doses of antiepileptic medications (i.e. dose changes within the last 3 months).
4. Patients with hypersensitivity to riluzole or any components of its formulation.
5. Patients with one or more of the following: HIV, Hepatitis B virus, Hepatitis C virus, hemophilia (bleeding problems, recent nose and brain injuries), abnormal blood pressure (hypotension or hypertension), drug abuse, immunity disorder, major depressive episode or psychosis.
6. Patients unable to tolerate venipuncture procedures for blood sampling.
7. Patients receiving concomitant medications that specifically target the glutamate system (e.g. memantine, d-cycloserine), or decrease the elimination of riluzole (e.g. theophylline, quinolones), less than 30 days prior to the screening visit.
8. Patients actively enrolled in another intervention study.
9. Patients who are unable to swallow pills.
10. Patients who have elevated liver enzymes ≥ 3 times the normal amount before the study begins.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 58 (Actual)
Dates: Start 2013-09; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Efficacy of riluzole vs. placebo on measures of social function | 12 weeks
  This will be measured by the Aberrant Behavior Checklist (ABC) - Lethargy / Social Withdrawal Subscale
Efficacy of riluzole vs. placebo on measures of repetitive behaviors | 12 weeks
  This will be measured by the Child Yale-Brown Obsessive Compulsive Scale (CY-BOCS)
Efficacy of riluzole vs. placebo on measures of repetitive behaviors | 12 weeks
  This will be measured by the Repetitive Behavior Scale (RBS-R)
Safety and tolerability of riluzole in children and adolescents with ASD | 12 Weeks
  This will be measured by the Safety Monitoring Uniform Report Form (SMURF)
Safety and tolerability of riluzole in children and adolescents with ASD | 12 Weeks
  This will be measured by the Clinical Global Impressions - Improvement Scale - Global (CGI-I-Global)

CONTACTS AND LOCATIONS:
Overall Officials: Evdokia Anagnostou, M.D., Principal Investigator — Holland Bloorview Kids Rehabilitation Hospital; Robert Nicolson, M.D., Principal Investigator — University of Western Ontario, Lawson Health Research Institute; Terry Bennett, M.D., Principal Investigator — McMaster University; Offord Centre for Child Studies
Locations (3):
- Canada (3):
  - Offord Centre for Child Studies, Hamilton, Ontario
  - Lawson Health Research Institute, London, Ontario
  - Holland Bloorview Kids Rehabilitation Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No